CLINICAL TRIAL: NCT06514287
Title: Telehealth Intervention for Performance of Activities in Daily Routines in Children and Adolescents With Disabilities
Brief Title: Telehealth Interventions for Daily Routine Activities in Children and Adolescents With Disabilities
Acronym: Telehealth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European University Miguel de Cervantes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI-DOC006-Telehealth
Record Dates: First submitted 2024-07-08; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Children With Physical Disabilities; Adolescents With Physical Disabilities
Keywords: children; adolescents; disability; physical therapy; participation; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individualized intervention (Other): It is a pragmatic intervention where three priorities were identified for physical activities in daily routines, considering the difficulty of the goal, the family's daily routines, opportunities for practice, and time available for practice. The therapist is a consultant, sharing information, educating, and instructing in ways that encouraged engagement of participants in the intervention process. The intervention plan was implemented via online consultation using WhatsApp text, audio, and video messaging for asynchronous and synchronous communication. The focus of intervention was incorporating practice of goals into daily activity routines.
  Interventions: Behavioral: Individualized intervention

INTERVENTIONS:
Behavioral: Individualized intervention — It is a pragmatic intervention where three priorities were identified for physical activities in daily routines, considering the difficulty of the goal, the family's daily routines, opportunities for practice, and time available for practice. The therapist is a consultant, sharing information, educating, and instructing in ways that encouraged engagement of participants in the intervention process. The intervention plan was implemented via online consultation using WhatsApp text, audio, and video messaging for asynchronous and synchronous communication. The focus of intervention was incorporating practice of goals into daily activity routines.

SUMMARY:
Performance of activities during daily routines is an important outcome of rehabilitation services for children and adolescents with physical disabilities, independent of their health condition or functional level. The aim of this study was to evaluate the effect of a telehealth intervention using WhatsApp text, audio, and video messaging on achievement of individualized goals for performance of activities in daily routines in children and adolescents with physical disabilities. The intervention is an eight-week participation-based intervention for children and adolescents with physical disabilities consisted of a goal-oriented, family-centred, collaborative, strength-based, ecological, and self-determined intervention.

DETAILED DESCRIPTION:
Performance of activities during daily routines is an important outcome of rehabilitation services for children and adolescents with physical disabilities, independent of their health condition or functional level. The International Classification of Functioning, Disability, and Health defines activity as whole-body actions and participation as involvement in life situations. Telehealth is a method of service delivery that might enable service providers and families to collaborate on goals for performance of activities during daily routines. The aim of this study was to evaluate the effect of a telehealth intervention using WhatsApp text, audio, and video messaging on achievement of individualized goals for performance of activities in daily routines in children and adolescents with physical disabilities.

The intervention is an eight-week participation-based intervention for children and adolescents with physical disabilities consisted of a goal-oriented, family-centred, collaborative, strength-based, ecological, and self-determined intervention. It is a pragmatic intervention where goals for physical activities in daily routines took into consideration the difficulty of the goal, the family's daily routines, opportunities for practice, and time available for practice. The therapist is a consultant, sharing information, educating, and instructing in ways that encouraged engagement of participants in the intervention process. There are two follow-ups: first after twelve weeks y the last two years later.

ELIGIBILITY:
Inclusion Criteria:

* Participants between five and 21 years old.
* Participants with a physical disability.
* Participants with the ability to walk with or without an assistive device.

Exclusion Criteria:

* Participants with orthopedic surgery within the past 6 months.
* Participants with a health condition limiting physical activity.
* Participants with contraindications to exercise.
* Participants unable to understand the instructions to complete the outcome measures.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2024-10-25 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | 0 week, 8 weeks, 20 weeks
  The COPM is an individualized outcome measure of a client's perception of their occupational performance. Occupational performance refers to an individual's experiences in performing activities in daily life. The parent or child identify their priorities for activities in daily living. After priorities are identified, each is rated for current performance and satisfaction with current performance on a scale of 1 (not able to do it / not satisfied at all) to 10 (able to do it extremely well / extremely satisfied). An increase of two or more points for is considered a clinically significant change.
Goal Attainment Scaling (GAS) | 0 week, 8 weeks, 20 weeks
  GAS is a standardized individualized outcome measure in which five measurable outcomes are specified for each goal. A score of -2 indicates the level of function at the start of intervention, 0 is the expected level of function, and +2 indicates a level of function that far exceeds the expected level of function following the intervention. The composite change score is expressed as a standardized T-score (mean = 50, standard deviation = 10). A T-score of 50 corresponds to achievement at the expected level.
Activity log | 8 weeks
  Participants were provided a sheet that listed the activities for each goal listed and asked to record the days and times activities were practiced.
Interviews to families | 8 weeks, 20 weeks, 124 weeks
  At post-intervention, short follow-up and long follow-up, participants were asked about the practice or their individualized goals, if the intervention was useful for them, and if the intervention empower them to plan new personal goals in the future and ask for help, when needed. The responses will be recorded.
Functional variables: physical activity levels with accelerometery | 0 week, 8 weeks, 20 weeks
  It is one of the most reliable techniques for recording and storing the amount and level of physical activity performed by each person in a given period of time, considering mainly light physical activity (LPA) and moderate to-vigorous activity (MVPA). The levels of physical activity of the participants will be recorded over a seven-day period using the GT3X+ accelerometer. The output from the ActiGraph will be provided in 'counts'.
Functional variables: physical activity levels with questionnaires | 0 week, 8 weeks, 20 weeks
  Physical activity levels are recorded using an PAQ-C PAQ-A Physical Activity Questionnaire for children and adolescents (PAQ-C and PAQ-A). They are self-administered questionnaires to measure physical activity levels in children aged approximately 8-14 years (PAQ-C) and adolescents aged approximately 14-20 years (PAQ-A).
Functional variables: gas consumption analysis | 0 week, 8 weeks, 20 weeks
  Changes in oxygen consumption (VO2) and carbon dioxide production (CO2).
Functional variables: Heart rate | 0 week, 8 weeks, 20 weeks
  Changes in heart rate, measured by a polar H10 Heart Rate Monitor with Chest Strap.
Clinical variables: Body composition | 0 week, 8 weeks, 20 weeks
  Changes in measurements by Body Mass Index (BMI), where weight and height will be combined to report it in kg/m^2.
Clinical variables: Bioelectrical Impedance Analysis | 0 week, 8 weeks, 20 weeks
  Changes in fat mass percentage.
Children's Assessment of Participation and Enjoyment (CAPE) | 0 week, 8 weeks, 20 weeks
  It is a tool designed to record how the child, with or without a disability, participates in 55 daily activities outside of school activities. It addresses the diversity (0- no practised, 1- practised) and intensity of the child's activity participation (scoring 1-7, where 1 is less to 7 more practice), with whom and where the activities are typically done (scoring form 1-5, 1 alone to 5 with others), and the child's enjoyment of the activities (scoring 1-5, 1- no enjoyment at all to 7- I love it).
Participation and Environment Measure for Children and Youth (PEM-CY) | 0 week, 8 weeks, 20 weeks
  It is a parent-reported tool that examines participation and environmental factors affecting child participation in three contexts: home, school, and community. Summary scores are calculated for frequency (average, 0-never to 7-daily), involvement (average, 1-minimally involved to 5-very involved), and perceived environmental support (percentage).
Muscle thickness of the vastus lateralis quadriceps with ultrasound | 0 week, 8 weeks, 20 weeks
  The thickness of the muscle (mm) will be recorded by performing longitudinal and transverse ultrasound images.
Pennation angle of the vastus lateralis quadriceps with ultrasound | 0 week, 8 weeks, 20 weeks
  The pennation angle (degree) of the muscle will be recorded by performing longitudinal and transverse ultrasound images.
Muscle strength | 0 week, 8 weeks, 20 weeks
  Measured by manual digital dynamometry of the quadriceps muscle groups.
Muscle strength measured by Five times sit to stand test (FTSTS) | 0 week, 8 weeks, 20 weeks
  This is a test to evaluate the functional strength of the lower extremities.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Santos Lozano, PhD, Principal Investigator — Universidad Europea Miguel de Cervantes
Locations (1):
- European University Miguel of Cervante, Valladolid, Castille and León, Spain

REFERENCES:
- [Result] Palisano RJ, Chiarello LA, King GA, Novak I, Stoner T, Fiss A. Participation-based therapy for children with physical disabilities. Disabil Rehabil. 2012;34(12):1041-52. doi: 10.3109/09638288.2011.628740. Epub 2011 Nov 14. PMID 22080765
- [Result] Organization, W. H., IFC: International Classification of Functioning, Disability and Health. 2001.
- [Derived] Matey-Rodriguez C, Pico M, Robles-Garcia V, Musso-Daury L, Santos-Lozano A, Palisano RJ. Collaborative Telehealth Intervention for Performance of Activities During Daily Routines by Children and Adolescents with Physical Disabilities: A Feasibility Study. Phys Occup Ther Pediatr. 2026 Jan 19:1-19. doi: 10.1080/01942638.2026.2618039. Online ahead of print. PMID 41555535